CLINICAL TRIAL: NCT05893407
Title: Quantification of Cerebral Perfusion at the Patient's Bedside When Performing Contrast-enhanced Ultrasound in Neurointensive Care Patients
Brief Title: Brain PERfusion Evaluation by Contrast-Enhanced UltraSound
Acronym: PerCEUS
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230489; 2023-A00939-36 (Other: IDRCB number)
Record Dates: First submitted 2023-05-29; First posted 2023-06-07 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Cerebral Hemorrhage; Subarachnoid Hemorrhage; Ischemic Stroke; Cerebrovascular Circulation; Perfusion
Keywords: Brain perfusion; Cerebral blood flow; Diagnostic imaging; Ultrasonography Doppler; Doppler ultrasound; Transcranial Doppler; Contrast enhanced ultrasound; Contrast-enhanced ultrasonography; Contrast ultrasound; Ultrasound perfusion imaging; Ultrasound contrast agent; Intra-cranial pressure; Intracerebral hematoma; Neurocritical care
MeSH Terms: conditions — Cerebral Hemorrhage; Subarachnoid Hemorrhage; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acute brain injuries when a contrast ultrasound imaging is requested by the physician: Contrast-enhanced ultrasound perfusion imaging (PerCEUS)
  Interventions: Diagnostic Test: Measuring contrast-enhanced ultrasound perfusion with phase inversion harmonic imaging

INTERVENTIONS:
Diagnostic Test: Measuring contrast-enhanced ultrasound perfusion with phase inversion harmonic imaging — Contrast-enhanced ultrasound perfusion imaging (PerCEUS) will be performed by a dedicated study team. The transcranial color duplex sonography will be performed with a 1-5 MHz dynamic sector array (S5-1) from a Philips Epiq 7 ultrasound machine (Philips Healthcare, Andover, MA). The field-of-view will be set to an imaging depth of 150 mm in a sector angle of 90°. The imaging plane will be then tilted to the diencephalic, in which the frontal horns of the side ventricles and the third ventricle serve as landmarks and where the anterior and posterior middle cerebral artery (MCA) territory and the basal ganglia (BG) as region of interest could be identified without artefacts from major vessels. High mechanical index bolus imaging will be performed from the sanest side of the head. Data acquisition of 45 seconds will be recorded immediately after the beginning of the contrast ultrasound imaging, using a mechanical index (MI) setting of 1.1 and a frame rate of 33 Hz.

SUMMARY:
The objective of the study is to assess brain tissue perfusion by contrast-enhanced ultrasound perfusion imaging (PerCEUS) in acute brain injuries. More precisely, it aims :

* to evaluate the heterogeneity of brain perfusion and thus diagnose brain tissue hypoperfusion with contrast-enhanced ultrasound.
* to correlate contrast-enhanced ultrasound with perfusion measurements by usual multimodal monitoring.

DETAILED DESCRIPTION:
The main aim is to evaluate the heterogeneity of brain perfusion, thus diagnosing brain tissue hypoperfusion with PerCEUS, then to correlate it with the usual multimodal monitoring.

Earlier after hospitalization in neurointensive care, when the study physician needs to realize a contrast ultrasound imaging and without delaying any emergency procedure, a PerCEUS will be performed in patients with an acute brain injury. After acquisition, data from PerCEUS will be transferred to an external evaluation unit and analysed offline, using commercially available software Qlab (Philips ®). According to the localization of acute brain injuries with magnetic resonance imaging (MRI) and/or computed tomography (CT), several regions-of-interest (ROI, at least three in each area) will be chosen :

* Area 1 : in the core of the lesion (supposed non perfused)
* Area 2 : just next to the lesion (supposed hypoperfused)
* Area 3 : in the saner hemisphere, symmetrically to area 2 each time it's possible (supposed well-perfused).

Every parameters of multimodal monitoring used at the moment of PerCEUS will be relieved :

* intracranial pressure (ICP), cerebral perfusion pressure (CPP), mean arterial pressure (MAP)
* mean flow velocity (MFV) by transcranial doppler (TCD)
* regional cerebral oxygen saturation (rSO2) by Near infrared spectroscopy (NIRS)
* jugular venous oximetry (SjvO2).

The actual PerCEUS measurement takes place at the bedside, is performed by the study physician, and takes about 5 minutes.

The trial duration per patient is 30 minutes, ending after 25 minutes of oversight

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Intensive care unit admission for acute brain injury
* Proven acute brain injury by CT and/or MRI
* Requiring a contrast ultrasound imaging
* Informed consent of patient or relative

Exclusion Criteria:

* Pregnancy
* Not sufficient temporal window
* Contraindications to Sonovue ® : acute coronary syndromes, severe ischemic heart disease (requiring revascularization), pulmonary arterial hypertension > 90 mmHg, right-left shunt, ARDS, dobutamine's use, known allergy or adverse reaction to Sonovue®
* Patient on State Medical Assistance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in neurosurgical intensive care in Lariboisière Hospital, Paris, with acute brain injuries
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the heterogeneity of brain perfusion by time-to-peak (TPI) measurement | 30 minutes after PerCEUS
  Comparison between time-to-peak (TPI) intensities measured in ROIs in each area by PerCEUS
Evaluation of the heterogeneity of brain perfusion by peak-intensities (PI) measurement | 30 minutes after PerCEUS
  Comparison between peak-intensities (PI) measured in ROIs in each area by PerCEUS

SECONDARY OUTCOMES:
Correlation between PerCEUS parameters and cerebral perfusion as assessed by ICP and MAP | 30 minutes after PerCEUS
  Correlations test between TPI/PI and ICP/CPP/MAP
Correlation between PerCEUS parameters and cerebral perfusion as assessed by TCD | 30 minutes after PerCEUS
  Correlations test between TPI/PI and MFV
Correlation between PerCEUS parameters and cerebral perfusion as assessed by NIRS | 30 minutes after PerCEUS
  orrelations test between TPI/PI and rSO2
Correlation between PerCEUS parameters and cerebral perfusion as assessed by SjvO2 | 30 minutes after PerCEUS
  Correlations test between TPI/PI and SjvO2

CONTACTS AND LOCATIONS:
Overall Officials: Romain BARTHELEMY, MD, Principal Investigator — AP-HP Lariboisière Hospital, Department of Anaesthesia and Intensive Care
Locations (1):
- Lariboisière Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eyding J, Krogias C, Wilkening W, Postert T. Detection of cerebral perfusion abnormalities in acute stroke using phase inversion harmonic imaging (PIHI): preliminary results. J Neurol Neurosurg Psychiatry. 2004 Jun;75(6):926-9. doi: 10.1136/jnnp.2003.026195. PMID 15146019
- [Background] Eyding J, Fung C, Niesen WD, Krogias C. Twenty Years of Cerebral Ultrasound Perfusion Imaging-Is the Best yet to Come? J Clin Med. 2020 Mar 17;9(3):816. doi: 10.3390/jcm9030816. PMID 32192077
- [Background] Vinke EJ, Kortenbout AJ, Eyding J, Slump CH, van der Hoeven JG, de Korte CL, Hoedemaekers CWE. Potential of Contrast-Enhanced Ultrasound as a Bedside Monitoring Technique in Cerebral Perfusion: a Systematic Review. Ultrasound Med Biol. 2017 Dec;43(12):2751-2757. doi: 10.1016/j.ultrasmedbio.2017.08.935. Epub 2017 Sep 28. PMID 28964614
- [Background] Fung C, Heiland DH, Reitmeir R, Niesen WD, Raabe A, Eyding J, Schnell O, Rolz R, Z Graggen WJ, Beck J. Ultrasound Perfusion Imaging for the Detection of Cerebral Hypoperfusion After Aneurysmal Subarachnoid Hemorrhage. Neurocrit Care. 2022 Aug;37(1):149-159. doi: 10.1007/s12028-022-01460-z. Epub 2022 Feb 24. PMID 35211837
- [Background] Bilotta F, Robba C, Santoro A, Delfini R, Rosa G, Agati L. Contrast-Enhanced Ultrasound Imaging in Detection of Changes in Cerebral Perfusion. Ultrasound Med Biol. 2016 Nov;42(11):2708-2716. doi: 10.1016/j.ultrasmedbio.2016.06.007. Epub 2016 Jul 27. PMID 27475927